CLINICAL TRIAL: NCT05826067
Title: Systematic Analysis of Bacterial Multidrug Tolerance in Longitudinal Isolates of Patients That Are Prone to Developing Urinary Tract Infections
Brief Title: Study of E. Coli Isolates From Recurrent Urinary Tract Infections
Acronym: Per-UTI
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Per-UTI
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Infections; Patients With Suprabubic Catheter; Patients With Nephrostomy Catheter
Keywords: Urinary tract infection; Escherichia coli
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with UTI or catheter (suprapubic, nephrostomy): Patients with urinary tract infection caused by E. coli, with or without neurological disorders or patients that are planned to undergo the insertion of a suprapubic or nephrostomy catheter.
  Interventions: Other: collection of bacterial strains

INTERVENTIONS:
Other: collection of bacterial strains — Urine (and blood) samples will be collected following SOC procedures for diagnostic purposes, at each visit of the patient (initial visit, follow up study or visit for new episode. For patients needing a catheter, urine sample will be collected before the insertion of the catheter, and before renewal of the catheter. Catheter tips will also be collected and sonicated to isolate bacteria. E. coli will be stored for analysis.

SUMMARY:
Prospective study aiming at collecting clinical Escherichia coli isolates from patients with recurrent urinary tract infection; samples to be collected during routine procedures.

DETAILED DESCRIPTION:
In a clinical context, persisters are of potential concern as they perpetuate chronic infections and enhance the development of antibiotic resistance. Novel therapeutic strategies to combat persisters are therefore highly needed. Most mechanistic studies on persistence to date deal with lab strains. The main goal of this project is to define principles of persistence and its evolution in natural strains of E. coli isolated from patients. Isolates will be collected as follows, from three types of patients corresponding to 3 different clinical situations where recurrent infection is likely

(A) Patients with urinary tract infection caused by E. coli, with or without neurological disorders.

First visit : for patients suspected for UTI, a first urine sample is collected (as part of the routine diagnosis procedure for this type of infection), before starting any antibiotic treatment. Likewise, a blood sample is taken to establish a possible concomitant sepsis if considered useful by the doctor. If the diagnosis of UTI is confirmed, informed consent will be obtained after explanation of the study by the investigator, making clear that the patient will be included only if E. coli is isolated from the urine. If the patient agrees to participate, the samples will be stored at -80°C for further analysis. Using a standardized questionnaire, a detailed medical history concerning recent UTIs and antibiotics taken by the patients is composed, possibly with the help of the family doctor of the patient if he/she does agree.

Next visits: If the patients come back for another episode (at least 2 weeks after the end of the treatment for the previous episode has been resolved), or for a control visit, data concerning their recent UTI history and antibiotic use will be collected using standardized questionnaires. A new urine sample will be collected. If the patients consult their GP for a new episode, they will be asked to fill the form with their GP and instruct the lab where the analysis of the new sample is done to send the strain to Saint Luc (cost will be covered). Written instruction will be provided.

IMPORTANT: The collection of urine samples for this study will not impede SOC. Samples are taken following the protocols used for patients with UTIs (and sepsis). The antibiotic regimen will not be adapted based on these results. When signing the informed consent, the patients will be informed that they will not personally benefit from the study but help scientific research.

(B-C) Patients that are planned to undergo the insertion of a suprapubic or nephrostomy catheter.

Visit 1 These patients are seen at the ward or consultation for a variety of non-UTI related problems. During this visit, informed consent is obtained and the study is explained by the investigator. Using a standardized questionnaire, a detailed medical history concerning recent UTIs and antibiotics taken by the patients is composed possibly with the help of the family doctor of the patient if he/she does agree. A first urine sample is collected.

Visit 2 (if not performed in visit 1) Insertion of the catheter and collection of a new urine sample (again, this is part of standard of care and not a study procedure).

Next visits Regular exchange of the catheter, every 6 weeks at the urology department. During these visits, patients are asked about their recent UTI history and any antibiotic use. Prior to the exchange, a urine sample is taken and the tip of the old catheter is collected (as per standard of care). Isolates from urine will be frozen and tips of catheter will be processed for biofilm disruption and freezing of bacteria.

IMPORTANT: The collection of urine samples for this study will not impede SOC. Samples are taken following the protocols used for patients with UTIs (and sepsis). The antibiotic regimen (if any) will not be adapted based on these results. When signing the informed consent, the patients will be informed that they will not personally benefit from the study but help scientific research.

Patients will be recruited over a two years period. For each patient, the duration of the participation will correspond (A) to each episode of UTI with sepsis over that period of time and (B-C) to the period during which a catheter remains in place over the study period.

Directly after collection, biofilms on catheter tips will be disrupted following in-house protocols For both urine samples and catheter tip biofilms, bacterial strains will be isolated by inoculating on selective agar plates (MacConkey, mannitol salt, cetrimide …), followed by aerobic incubation at 37°C for 24h. Bacterial isolates observed on the selective media plates will be aseptically subcultured onto freshly prepared media plates and subjected to identification. For patients suffering from recurrent UTIs, the investigators expect to find mainly Escherichia coli while for patients with a suprapubic catheter the investigators expect mainly E. coli, as well as Pseudomonas aeruginosa, Proteus mirabilis and Klebsiella pneumoniae strains. Only E. coli will be stored for the study.

Isolates will then be transferred to research lab of the sponsor for further molecular analysis (determination of persister character in the presence of antibiotic, WGS, essentially).

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for urinary tract infection, with or without neurological disorders (spina bifida, MS, paraplegic patients) or ambulatory patients diagnosed with a urinary tract infection when the identified causative agent is E. coli
* patients who have or are planned to undergo the insertion of a suprapubic catheter
* patients who have or are planned to undergo the insertion a nephrostomy catheter

Exclusion Criteria: patients

* refusing the planned treatment
* with therapy compliance
* pregnant women
* who do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ambulatory patients coming to the hospital for a visit to the nephrology department or patients hospitalized in nephrology department
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
collection of longitudinal E. coli to be used for fundamental research | collection till the end of 2024
  To collect longitudinal bacterial isolates of E. coli and to record clinical data for fundamental research about patients that are prone to developing urinary tract infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaban NQ, Helaine S, Lewis K, Ackermann M, Aldridge B, Andersson DI, Brynildsen MP, Bumann D, Camilli A, Collins JJ, Dehio C, Fortune S, Ghigo JM, Hardt WD, Harms A, Heinemann M, Hung DT, Jenal U, Levin BR, Michiels J, Storz G, Tan MW, Tenson T, Van Melderen L, Zinkernagel A. Definitions and guidelines for research on antibiotic persistence. Nat Rev Microbiol. 2019 Jul;17(7):441-448. doi: 10.1038/s41579-019-0196-3. PMID 30980069